CLINICAL TRIAL: NCT07183176
Title: Treatment of Acute Low Back Pain With Transcutaneous Electrical Neurostimulation at the Emergency Department: a Randomized Controlled Trial
Acronym: TENS BACK PAIN
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 202418NOV504
Record Dates: First submitted 2025-09-12; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Acute Back Pain; Emergency Department Patient

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: If the patient is eligible and agrees to take part in the study:
  Stage 1: The doctor "investigator 1" carries out randomisation
  * Randomisation will be carried out by statistical support via the REDCap project.
  * The patient will be assigned to one of two groups:
    1. The intervention group: called the REAL TENS group (R- TENS)
    2. The control group: called the FAKE TENS group (F-TENS)
       Step 2: The doctor "investigator 1" will place the TENS on the painful area identified by the patient, following the model proposed in appendix 1.
       Step 3: The doctor "investigator 1" will explain to patients in both groups that they may feel a slight tingling sensation or no sensation at all.
       Step 4: The doctor "investigator 1" will make the following settings on the TENS:
  * For the interventional group (REAL TENS) a combined setting will be used:
    1. Tens Burst (P2) at 2Hz and 180 µs with an action on muscle pain.
    2. Tens gate control (P9) at 100 Hz and 250 µs with an action focused on nociceptive
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- REAL TENS group (R- TENS) (Experimental): The intervention group. Chattanooga CEFAR Tens
  Interventions: Device: Chattanooga CEFAR Tens
- FAKE TENS group (F-TENS) (Placebo Comparator): The control group
  Interventions: Device: Chattanooga CEFAR Tens

INTERVENTIONS:
Device: Chattanooga CEFAR Tens — * The patient will be assigned to one of two groups:
    1. The intervention group: called the REAL TENS group (R- TENS)
    2. The control group: called the FAKE TENS group (F-TENS)
       Step 2: The doctor "investigator 1" will place the TENS on the painful area identified by the patient, following the model proposed in appendix 1.
       Step 3: The doctor "investigator 1" will explain to patients in both groups that they may feel a slight tingling sensation or no sensation at all.
       Step 4: The doctor "investigator 1" will make the following settings on the TENS:
  * For the interventional group (REAL TENS) a combined setting will be used:
    1. Tens Burst (P2) at 2Hz and 180 µs with an action on muscle pain.
    2. Tens gate control (P9) at 100 Hz and 250 µs with an action focused on nociceptive pain.
  * For the control group (FAKE TENS), the doctor will not make any "real" adjustments.
  The patient will not be able to see the settings made by the doctor "investigator 1".
  Stage 5: The doctor "investigator
  Other Names: FAKE Tens

SUMMARY:
Acute low back pain is a frequent cause of emergency department admissions (4.39% [95% CI: 3.67-5.18])1. Drug therapeutic options are limited and ineffective. Paracetamol and opioids are no better than placebo for acute low-back pain 2,3. Only NSAIDs and muscle relaxants have a slightly beneficial effect on pain, but muscle relaxants have an unfavorable risk-benefit balance.2 In this situation, it is necessary to turn to new non-drug therapeutic options to relieve pain of these patients. Transcutaneous electrical nerve stimulation (TENS) is a non-drug therapy that involves applying an electrical current through the skin. Through one or two pairs of electrodes stuck to the skin, TENS delivers painless, low-intensity electrical impulses to a painful area or a nerve pathway.

TENS acts by selectively activating large-diameter non-nociceptive afferent fibers to induce segmental analgesia4. In addition, TENS increases the concentration of endorphins in the bloodstream and cerebrospinal fluid5.

The use of TENS has been studied mainly in chronic low-back pain. A 2007 Cochrane systematic review concluded that TENS appears to reduce pain and improve range of motion for subjects with chronic low back pain6.

The use of TENS in emergency departments has been little studied. A 2018 pilot study of 110 patients admitted to the emergency department with acute or chronic pain observed a reduction in pain (from an average of 8.50 on the numerical pain scale [EN] [7.52 - 9.48] to 4.67 [3.51 - 5.89]) after TENS use and functional improvement in 83% of patients7.

The Gulacti study, carried out in 2022, investigated the use of TENS to treat pain of patients admitted to the emergency department with a renal colic attack : the mean reduction in VAS score at 15 and 30 minutes was significantly greater for the TENS group than for the placebo group (mean reduction in VAS score at 15 minutes was 33.3 ± 17.6 (95% CI : 28.3 to 38.3) for the TENS group and 14.9 ± 11.6 (95% CI: 11.6 to 18.2) for the placebo group [mean difference: 18.4 (95% CI: 12.5 to 24.4, P < 0.0001)]. The mean reduction in VAS score after 30 minutes was 63.7 ± 21.1 (95% CI: 57.7 to 69.7) for the TENS group and 14.9 ± 16.2 (95% CI: 19.5 to 10.3) for the placebo group (mean difference: 48.8, 95% CI: 41.4 to 56.3, P < 0.0001)8.

A single study of 76 patients focused on acute low-back pain during patient transport to emergency departments. The authors recorded a significant reduction (p= 0.01) in pain during transport of the TENS group (79.2 ± 6.5 mm VAS to 48.9 ± 8.2 0 mm VAS), while pain scores remained unchanged for the placebo group (75.9 ± 16.4 mm VAS and 77.1 ± 11.2 mm VAS)9.

To our knowledge, there is no high-quality study of TENS versus placebo for acute low back pain of patients admitted to an emergency department.

1. Primary objective:

   Study the analgesic efficacy of TENS compared to placebo in the treatment of acute low back pain at the emergency department.
2. Secondary objective:

1. Compare the number of patients who will show a > 50% reduction of their initial pain.

2. Compare the number of patients requiring rescue treatment. 3. Compare the occurrence of side effects among groups. 4. Compare patient satisfaction after 30 minutes. 5. Compare patient comfort level after 30 minutes.

Main criterion:

Comparison of the proportion of patients with >30% reduction of initial pain after 30 minutes of treatment

Secondary criterion:

1. Proportion of patients with > 50% reduction of their initial pain after 30 minutes of treatment.
2. Proportion of patients requiring morphine titration for pain relief.
3. The rate of side-effects associated with the use of TENS.
4. The level of satisfaction measured by numerical satisfaction scale ranging from 0 (not at all satisfied) to 10 (extremely satisfied) EN. A patient will be considered very satisfied if he/she presents a satisfaction level ≥ 8.
5. The level of comfort will be assessed by a comfort scale ranging from 0 (not at all comfortable) to 10 (very comfortable patient).

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to the emergency department and aged over 18 years with pain (EN > 3) related to acute low back pain.

The lumbar region is defined as the anatomical area between the costal margin and the gluteal fold.

Acute low back pain is defined by the World Health Organisation, and by part of the literature, as a low back pain that appeared less than 6 weeks ago.

Exclusion Criteria:

Refusal to participate in study, refusal to sign informed consent

* Consent is impossible to obtain (cognitive impairment, language barrier, etc.)
* Patients with low back pain lasting more than > 6 weeks
* Pregnant women
* Patient requiring immediate medical attention (vital distress).
* Patient already treated with a TENS
* Patient with a body temperature > 38°C
* Patient known to have a spinal infection
* Lumbar pain linked to trauma
* Patient with known systemic or spinal rheumatological disease
* Patient with a known systemic inflammatory disease
* A patient with a known chronic pain condition such as fibromyalgia
* Patient with pain radiating into the lower limb along the course of one of the following nerves (L3-L4-L5- S1)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2026-09-15 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
Comparison of the proportion of patients with >30% reduction of initial pain after 30 minutes of treatment | 30 minutes

SECONDARY OUTCOMES:
Proportion of patients with > 50% reduction of their initial pain after 30 minutes of treatment. | 30 minutes
Proportion of patients requiring morphine titration for pain relief. | 30 minutes
The rate of side-effects associated with the use of TENS. | 30 minutes
The level of satisfaction measured by numerical satisfaction scale ranging from 0 (not at all satisfied) to 10 (extremely satisfied) EN. A patient will be considered very satisfied if he/she presents a satisfaction level ≥ 8. | 30 minutes
The level of comfort will be assessed by a comfort scale ranging from 0 (not at all comfortable) to 10 (very comfortable patient). | 30 minutes

IPD SHARING:
Plan to Share IPD: Undecided